CLINICAL TRIAL: NCT01948960
Title: Influence of Exceptional Patient Characteristics on Everolimus Exposure
Acronym: INPRES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UMCNONCO201301
Record Dates: First submitted 2013-09-13; First posted 2013-09-24 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2017-10

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; everolimus; pharmacokinetics; elderly patients; obese patients
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care (No Intervention): everolimus dose is continued independently of everolimus AUC
- everolimus dose escalation (Active Comparator): patients with an AUC below mean will have dose escalation of everolimus based on their AUC
  Interventions: Drug: everolimus dose escalation

INTERVENTIONS:
Drug: everolimus dose escalation — patients with an AUC below mean will have dose escalation of everolimus based on their AUC
  Arms: everolimus dose escalation

SUMMARY:
A study to determine whether everolimus pharmacokinetics in elderly and obese patients is different compared to control patients.

Furthermore the investigators will investigate the relation between metabolic response assessed with [18F] Fluorodeoxyglucose-Positron Emission Tomography (FDG-PET) and everolimus exposure and clinical benefit.

The investigators will explore whether dose escalation in patients who are hypothetically underexposed will result in an increase in metabolic response.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 years of age) with metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy.
* Histological or cytological confirmation of estrogen-receptor positive (ER+) breast cancer
* Postmenopausal women
* Radiological or clinical evidence of recurrence or progression on last systemic therapy prior to enrollment.
* Progression following a non-steroidal aromatase inhibitor
* Falling into one of the following categories

  * elderly patients (age ≥ 70 years and BMI < 30 kg/m2); or
  * obese patients (BMI ≥ 30 kg/m2 and age < 70 years); or
  * control patients (BMI < 30 kg/m2 and age < 70 years);
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 x ULN
* Adequate renal function: calculated creatinine clearance, as estimated by GFR using the MDRD formula, is ≥ 30ml/min/1.73m2
* Performance status ECOG 0 - 2 (Karnofsky index: 60 - 100)
* Patient is willing and able to sign the Informed Consent Form prior to screening evaluations

Exclusion Criteria:

* Patients aged ≥ 70 years AND BMI ≥ 30 kg/m2
* HER2-overexpressing patients by local laboratory testing (IHC 3+ staining or in situ hybridization positive).
* Previous treatment with exemestane or mTOR inhibitors. Except for the treatment with exemestane in the adjuvant setting.
* Known hypersensitivity to mTOR inhibitors, e.g. sirolimus (rapamycin).
* Patients with a known history of HIV seropositivity.
* Any severe and / or uncontrolled medical conditions such as:

  * Unstable angina pectoris, serious uncontrolled cardiac arrhythmia
  * Patients with severe hepatic impairment (Child-Pugh A/B/C)
  * Uncontrolled diabetes mellitus
  * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
* Patients who test positive for hepatitis B or C
* Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A within the last 5 days prior to enrollment
* History of non-compliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-08; Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
everolimus AUC | day 14 after start treatment
  The primary aim is to show a difference in everolimus exposure (AUC0-24hr) of at least 25% in elderly patients (≥70 years) and obese patients (BMI ≥ 30 kg/m2) compared to the control group (≤ 70 years; BMI ≤ 30 kg/m2), after reaching steady state everolimus pharmacokinetics (day 14, but at least after 7 days of everolimus therapy).

SECONDARY OUTCOMES:
correlation between early metabolic response and PFS | within 90 days after start of treatment
  To explore and calculate the predictive value of early metabolic response assessment with clinical benefit (PFS defined as disease progression according to RECIST version 1.1 or death, whichever occurs first) as primary outcome measure.
  Metabolic response is defined as fractional change (ΔSUV and ΔTLG), comparing the third en second scan with the baseline scan.
correlation between early metabolic response and AUC | 15 days after start of treatment
  To quantify the correlation between early metabolic response and everolimus exposure (AUC0-24hr) on steady-state pharmacokinetics.
  Metabolic response is defined as fractional change (ΔSUV and ΔTLG), comparing the third en second scan with the baseline scan.
effect dose escalation on metabolic respons | within 36 days after start of treatment
  To explore, quantify and describe whether dose escalation in patients who are hypothetically underexposed will result in an increase in metabolic response.
  Metabolic response is defined as fractional change (ΔSUV and ΔTLG), comparing the third en second scan with the baseline scan.
correlation between AUC and frequency of adverse event | 4 months after start of treatment
  To explore, quantify and describe the correlation between everolimus exposure and the frequency of adverse events as graded with CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Carla van Herpen, MD, PhD, Principal Investigator — Radboud university medical center, department of medical oncology; Nielka van Erp, PharmD, PhD, Principal Investigator — Radboud university medical center, department of Pharmacy
Locations (7):
- Netherlands (7):
  - Maasziekenhuis Pantein, Boxmeer
  - Spaarne Gasthuis, Hoofddorp
  - Maastricht University Medical Center, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - Radboud university medical center, Nijmegen
  - Bernhoven Ziekenhuis, Uden
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] Willemsen AECAB, de Geus-Oei LF, de Boer M, Tol J, Kamm Y, de Jong PC, Jonker MA, Vos AH, Grootjans W, de Groot JWB, Mulder SF, Aarntzen EHJG, Gerritsen WR, van Herpen CML, van Erp NP. Everolimus Exposure and Early Metabolic Response as Predictors of Treatment Outcomes in Breast Cancer Patients Treated with Everolimus and Exemestane. Target Oncol. 2018 Oct;13(5):641-648. doi: 10.1007/s11523-018-0596-8. PMID 30259313
- See also: Everolimus Exposure and Early Metabolic Response as Predictors of Treatment Outcomes in Breast Cancer Patients Treated with Everolimus and Exemestane — https://www.ncbi.nlm.nih.gov/pubmed/30259313